CLINICAL TRIAL: NCT04386395
Title: Whole Blood Immune Cells Characterization in Critically Ill COVID-19 Patients: A Prospective Study
Brief Title: Immune Changes in Severe COVID-19 Pulmonary Infections
Acronym: COVIDIMM
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: CHRU NANCY : 2020PI080_1
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2020-12

CONDITIONS: SARS-CoV-2; Immune System Disorder
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immuno Cohort: COVID-19 confirmed ICU patients, sedated and ventilated, sequential characterization of circulating immune cells over their ICU stay. Every 2 to 3 days, fresh whole blood aliquots from routine blood counts were processed on a Flow Cytometer (Beckman Coulter) to determine immune cells subpopulations
- Cortico Cohort: COVID-19 confirmed ICU patients, sedated and ventilated, sequential characterization of circulating immune cells over their ICU stay. According to RECOVERY study, early routine administration of dexamethasone 6 mg/day over 10 days. Every 2 to 3 days, fresh whole blood aliquots from routine blood counts were processed on a Flow Cytometer (Beckman Coulter) to determine immune cells subpopulations

SUMMARY:
SARS-CoV-2 outbreak causes a spectrum of clinical patterns that varies from asymptomatic infection to mildly symptomatic manifestations and more-severe forms that need intensive care. Until now, the immune response to SARS-CoV-2 virus infection has been poorly reported to help decision for immune modulation therapies. As a consequence, trials have been designed to test both anti-inflammatory molecules as steroids or anti-bodies against IL-6, and others proposing to "boost" immunity with interferon beta based on similar inclusion criteria.

The immune response to infective agents including viruses may have a complex time evolution with early and late phases corresponding to different patterns, oscillating between pro-inflammation and immune-depression. The potential window to improve outcome in COVID-19 by therapeutic intervention aimed at a fine tuning between immune toxicity and immunodepression requires a longitudinal assessment during the course of illness, especially for the patients who develop acute respiratory failure. Immune monitoring of both innate and adaptive immunity would then be essential to appropriately design clinical trials.

The whole blood cells evaluation was recorded according to the time intervals between the onset of symptoms and the sampling after ICU admission. Patients' care was standardized, especially with regard to ventilation, sedation, and antimicrobial treatment.

In this study the investigators prospectively perform a longitudinal study of both innate and adaptive immunity on patients admitted to ICU for an COVID-19 related acute respiratory failure. The data will be analyzed in reference to the onset of initial symptoms and also to the admission in ICU.

The primary end point is the evolution of the characterization of monocytes and their subsets in term of number and expression of HLA-DR. A similar approach is used for lymphocytes and their subtypes with in addition, an ex vivo testing of their capabilities to be stimulated by SARS-CoV-2 viral proteins in term of TNFalpha, INFgamma, and IL1beta production.

The secondary end-point was to test the association with outcomes and other non-specific markers of inflammation as CRP (C reactive protein), PCT (procalcitonin), DDimers and ferritin.

DETAILED DESCRIPTION:
The most severe form of COVID-19 treated in intensive care for acute respiratory failure may have a poor prognosis. Both the level of IL-6 and the severity of the lymphopenia have been associated to the poor prognosis. Better knowledge of the time evolution of the circulating immune cells subpopulations and functions will help to best tailor the treatment: anti-inflammatory strategy at the initial phase might be rapidly shifted to immune stimulation when immunodepression is diagnosed.

It is then essential to assess the patients' immune status using flowcytometry methods to characterize both innate and adaptive immunity of the whole blood circulating immune peripheral blood mononuclear cells (PBMC). After cell staining with the adequate cell markers, the flowcytometry (NAVIOS® Flow Cytometer (Beckman Coulter) allowed to analyze the number and the function of the cells with an adequate gating strategy and the Kaluza® software v2.1 (Beckman Coulter). The data were then grouped by time intervals referring to the onset of symptoms and also to the ICU admission. The trend for innate immunity (monocytes number and subpopulations, HLA-DR expression) and for adaptive immunity (lymphocytes and subpopulations) will be analyzed. Since it is unknown if whole blood CD3/CD4 and CD3/CD8 lymphocytes elicit an "exhaustion" pattern and/or an abnormal response, an ex vivo testing of their reactivity for SARS-CoV-2 viral proteins will be performed. This test of polyfunctionality will characterize the intracellular cytokine expression (IL-1 beta, TNFalpha, and INFgamma) both for CD4 and CD8 T cells.

ELIGIBILITY:
Inclusion Criteria: confirmed COVID-19

* a positive RT- PCR,
* a highly suggestive thoracic CTScan,
* severe hypoxemia

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 ICU patients, sedated and mechanically ventilated within the 48 hrs of admission for the first sampling, and monitored all over their ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in monocytes HLA-DR expression | through ICU stay, an average of 30 days
  circulating immune cell characterization
Changes in lymphocytes subpopulations numbers | through ICU stay, an average of 30 days
  circulating immune cell characterization
Changes in monocytes number | through ICU stay, an average of 30 days
  circulating immune cell characterization

SECONDARY OUTCOMES:
TNFalpha level | 4 hours
  stimulation by SARS-CoV-2 viral proteins
INFgamma level | 4 hours
  stimulation by SARS-CoV-2 viral proteins
IL1beta level | 4 hours
  stimulation by SARS-CoV-2 viral proteins
SOFA score | through ICU stay, an average of 30 days
  Sequential Organ dysfunction assessement, ranging from 0 (better) to 24 (worst) outcome
number of recorded deaths | through study completion, an average of 6 months
  mortality
presence of pneumonia | through ICU stay, an average of 30 days
  infectious complications
presence of bacteremia | through ICU stay, an average of 30 days
  infectious complications
presence of urinary tract infection | through ICU stay, an average of 30 days
  infectious complications
C reactive protein | through ICU stay, an average of 30 days
  inflammation marker
D Dimers | through ICU stay, an average of 30 days
  inflammation marker

CONTACTS AND LOCATIONS:
Overall Officials: MARIE REINE LOSSER, MD, PhD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Centre Hospitalier Universitaire NANCY, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Tan L, Wang Q, Zhang D, Ding J, Huang Q, Tang YQ, Wang Q, Miao H. Lymphopenia predicts disease severity of COVID-19: a descriptive and predictive study. Signal Transduct Target Ther. 2020 Mar 27;5(1):33. doi: 10.1038/s41392-020-0148-4. No abstract available. PMID 32296069
- [Background] Payen D, Faivre V, Miatello J, Leentjens J, Brumpt C, Tissieres P, Dupuis C, Pickkers P, Lukaszewicz AC. Multicentric experience with interferon gamma therapy in sepsis induced immunosuppression. A case series. BMC Infect Dis. 2019 Nov 5;19(1):931. doi: 10.1186/s12879-019-4526-x. PMID 31690258
- [Background] Ziegler-Heitbrock L, Ancuta P, Crowe S, Dalod M, Grau V, Hart DN, Leenen PJ, Liu YJ, MacPherson G, Randolph GJ, Scherberich J, Schmitz J, Shortman K, Sozzani S, Strobl H, Zembala M, Austyn JM, Lutz MB. Nomenclature of monocytes and dendritic cells in blood. Blood. 2010 Oct 21;116(16):e74-80. doi: 10.1182/blood-2010-02-258558. Epub 2010 Jul 13. PMID 20628149
- [Background] Hotchkiss RS, Monneret G, Payen D. Sepsis-induced immunosuppression: from cellular dysfunctions to immunotherapy. Nat Rev Immunol. 2013 Dec;13(12):862-74. doi: 10.1038/nri3552. Epub 2013 Nov 15. PMID 24232462
- [Background] Alattar R, Ibrahim TBH, Shaar SH, Abdalla S, Shukri K, Daghfal JN, Khatib MY, Aboukamar M, Abukhattab M, Alsoub HA, Almaslamani MA, Omrani AS. Tocilizumab for the treatment of severe coronavirus disease 2019. J Med Virol. 2020 Oct;92(10):2042-2049. doi: 10.1002/jmv.25964. Epub 2020 May 10. PMID 32369191
- [Background] Payen D, Cravat M, Maadadi H, Didelot C, Prosic L, Dupuis C, Losser MR, De Carvalho Bittencourt M. A Longitudinal Study of Immune Cells in Severe COVID-19 Patients. Front Immunol. 2020 Oct 23;11:580250. doi: 10.3389/fimmu.2020.580250. eCollection 2020. PMID 33178207